CLINICAL TRIAL: NCT07025941
Title: Impact of Comprehensive Rehabilitation Nursing Combined With Refined Airway Management and Nutritional Support on Prognosis and Care Delivery Models in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taizhou Hospital of Traditional Chinese Medicine (Other Government)
Responsible Party: Principal Investigator, Peibei zhang, Principal Investigator, Taizhou Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20240511
Record Dates: First submitted 2025-06-09; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Critically Ill Patients; Nutritional Support; Pulmonary Infections; Gastrointestinal Bleeding; Acute Kidney Injury (AKI)
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Acute Kidney Injury

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other)
  Interventions: Other: Standard Critical Care Nursing Protocol
- intervention group (Experimental)
  Interventions: Behavioral: ICU-PRO Nursing Protocol (Integrated Critical Care Protocol for Rehabilitation Outcomes)

INTERVENTIONS:
Other: Standard Critical Care Nursing Protocol — The Standard Critical Care Nursing Protocol encompasses evidence-based, routine nursing practices for critically ill patients in the intensive care unit (ICU). This protocol serves as the control intervention in comparative studies evaluating novel nursing strategies.
  Key Components:
  Basic Physiological Monitoring:
  Continuous assessment of vital signs (heart rate, blood pressure, respiratory rate, SpO₂).
  Strict intake/output monitoring and electrolyte balance management.
  Airway Management:
  Standard oxygen therapy (nasal cannula, face mask) or mechanical ventilation as prescribed.
  Scheduled suctioning, positional changes, and oral care (every 4-6 hours).
  Infection Prevention:
  Aseptic techniques for invasive procedures (e.g., central line care, urinary catheter management).
  Ventilator-associated pneumonia (VAP) bundle compliance (e.g., head-of-bed elevation, sedation vacations).
  Mobility & Skin Integrity:
  Passive range-of-motion exercises for immobilized patients (2×/day).
  Pr
  Arms: control group
Behavioral: ICU-PRO Nursing Protocol (Integrated Critical Care Protocol for Rehabilitation Outcomes) — The intervention group received a standardized 14-day nursing protocol combining three evidence-based components:
  Comprehensive Rehabilitation Nursing:
  Early mobilization protocol with passive/active exercises (3-4 sessions/day)
  Respiratory training using incentive spirometry (Triflo II® devices)
  Swallowing rehabilitation with VitalStim® electrical stimulation
  Refined Airway Management:
  Humidification via Fisher & Paykel® MR850 systems (33-44 mg/L)
  Closed suction systems (Ballard® Trach Care) with strict aseptic technique
  Oral care with 0.12% chlorhexidine solution (Peridex®) 4×/day
  Nutritional Support:
  Enteral feeding using Abbott Nutrition® formulas
  Parenteral nutrition via Baxter®/Fresenius Kabi® solutions
  Gastric residual monitoring with Kangaroo™ feeding pumps
  Key Features:
  Implemented by specialized ICU nurses, respiratory therapists, and dietitians
  Daily monitoring using Philips® IntelliVue patient monitors
  Protocol adjustments based on weekly APACHE II scoring
  Arms: intervention group

SUMMARY:
This combined intervention protocol effectively improves the prognosis of critically ill patients and optimizes nursing management models

DETAILED DESCRIPTION:
To investigate the impact of comprehensive rehabilitation nursing combined with refined airway management and nutritional support on the prognosis of critically ill patients and nursing management models, and to develop a new care management protocol. Critically ill patients were divided into a control group (routine nursing) and an intervention group (comprehensive rehabilitation nursing combined with refined airway management and nutritional support). Complications such as pulmonary infection and gastrointestinal bleeding, as well as clinical indicators including oxygen saturation (SpO₂), mechanical ventilation time (MVT), and length of stay (LOS), were compared between the two groups. Logistic regression and XGBoost models were constructed to analyze key influencing factors.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of ICU admission standards with critical illness confirmed by attending physicians or senior specialists
* Age ≥ 18 years
* Stable vital signs:

Systolic blood pressure ≥ 90 mmHg and ≤ 180 mmHg

Heart rate ≤ 120 beats/min

Oxygen saturation (SpO₂) ≥ 85% under ≤ 60% fraction of inspired oxygen (FiO₂)

* Intact or tolerable gastrointestinal (GI) function for enteral nutrition
* Informed consent from both patients and families Exclusion Criteria:(1)
* Terminal malignancies
* Brain death
* Irreversible organ failure (e.g., end-stage cirrhosis, advanced heart failure)
* Comorbidities potentially confounding study outcomes
* Contraindications to interventions (e.g., laryngeal edema, complete intestinal obstruction)
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-23 (Actual)

PRIMARY OUTCOMES:
ICU Length of Stay (LOS) | From randomization to ICU discharge, up to 60 days
  Calendar days from ICU admission to discharge criteria met (APACHE II score ≤10, hemodynamic stability for ≥24h).

SECONDARY OUTCOMES:
Incidence of Pulmonary Infections | From ICU admission to 48 hours post-extubation or 14-day intervention period
  Rate of ventilator-associated pneumonia (VAP) and other pulmonary infections confirmed by clinical criteria (temperature >38°C or <36°C, purulent secretions, leukocytosis >10×10⁹/L or leukopenia <4×10⁹/L) plus microbiological evidence from sputum/BALF cultures.

OTHER OUTCOMES:
Protocol Adherence Rate | Daily during 14-day intervention
  Percentage completion of scheduled:
  1. Rehabilitation sessions (≥80% sessions completed)
  2. Airway care procedures (per protocol)
  3. Nutritional targets (≥90% calorie/protein goals)

CONTACTS AND LOCATIONS:
Locations (1):
- Taizhou Hospital of Traditional Chinese Medicine, Taizhou, Jiangsu, China